CLINICAL TRIAL: NCT01049919
Title: MarrowStim PAD Kit for the Treatment of Critical Limb Ischemia (CLI) in Subjects With Severe Peripheral Arterial Disease (PAD)
Brief Title: Safety and Efficacy Study of Autologous Concentrated Bone Marrow Aspirate (cBMA) for Critical Limb Ischemia (CLI)
Acronym: MOBILE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary endpoint not met, remaining long-term follow-up not needed.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB-IDE 13996; BBIO.CR.CT002 (Other: Biomet)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: Critical Limb Ischemia; Peripheral Arterial Disease; Peripheral Vascular Disease; CLI; PAD; PVD; Angiogenesis; Stem Cells; Cell Therapy; Limb Salvage; Amputation; Leg Pain
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Concentrated bone marrow aspirate (cBMA) (Experimental): Collection of autologous bone marrow aspirate and point-of-care concentration using the bone marrow concentration device, followed by intramuscular injection of concentrated bone marrow aspirate (cBMA) into the affected limb
  Interventions: Device: Bone marrow concentration device
- Placebo control (sham) (Sham Comparator): Placebo procedure (sham) consists of simulated bone marrow aspiration followed by simulated intramuscular injections into the affected limb
  Interventions: Procedure: Placebo procedure (sham)

INTERVENTIONS:
Device: Bone marrow concentration device — Concentration of autologous bone marrow aspirate for intramuscular delivery to affected limb
  Other Names: Bone marrow concentrate; Bone marrow mononuclear cells; MarrowStim
  Arms: Concentrated bone marrow aspirate (cBMA)
Procedure: Placebo procedure (sham) — Sham bone marrow aspiration, sham delivery to affected limb
  Arms: Placebo control (sham)

SUMMARY:
This trial will evaluate the safety and efficacy of concentrated bone marrow aspirate (cBMA) to prevent or delay major amputation and/or death in subjects with critical limb ischemia (CLI) due to severe peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo controlled, multicenter trial intended for subjects with critical limb ischemia (CLI) that are unsuitable for revascularization. The investigational treatment utilizes autologous concentrated bone marrow aspirate (cBMA) at the point of care. The bone marrow aspirate is obtained from the subject's hip, concentrated with a bone marrow concentration device, and delivered intramuscularly to the affected limb. Subjects meeting the inclusion/exclusion criteria will be randomized to receive either the investigational treatment (cBMA) or a placebo control (sham treatment).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral lower extremity ischemia due to advanced peripheral arterial disease
* Unsuitable for revascularization
* Minor tissue loss (Rutherford Category 5) or ischemic rest pain (Rutherford Category 4) with ABI ≤ 0.6, or TBI ≤ 0.4, or TcPO2 ≤ 50 mm Hg
* Competent to give consent
* No current malignancy or history of previous malignancy within the last five years, with the exception of adequately treated non-melanoma skin cancer (evidence of standard preventative cancer screenings required)

Exclusion Criteria:

* Major tissue loss (Rutherford Category 6)
* Diabetics on oral or insulin therapy with uncontrolled or untreated proliferative retinopathy (evidence of retinal exam required)
* Poorly controlled diabetes mellitus with HbA1C > 10% (evidence of HbA1C test required)
* Uncompensated congestive heart failure (New York Heart Association Class IV) and/or other conditions that preclude general anesthesia
* Myocardial infarction or stroke within last 90 days
* Elevated liver function tests (AST or ALT more than twice normal upper limit)
* Renal disease (creatinine > 2.5 mg/dl) or chronic hemodialysis
* White blood cell count < 3,000/µL or > 15,000/µL, platelet count < 100,000/µL, or hematocrit < 32%
* Topical growth hormone therapy within last 90 days, or injected growth hormone therapy within last 180 days
* Disease of central nervous system and/or other conditions that impair cognitive function
* Two or more episodes of pulmonary embolus with a documented DVT in index leg or history of DVT in index leg without evidence of clot resolution
* Current infection of index leg
* Pregnant women (negative urine pregnancy test required)
* Lower extremity venous disease with pitting edema in index leg
* Recent history (in the 6 months prior to screening) of bone marrow disease or treatment with any medication or procedure which adversely affects the bone marrow and would prohibit transplantation
* Current osteomyelitis in index leg
* Existing HIV diagnosis
* Organ transplant recipients
* Known terminal disease process with life expectancy less than one year
* Severe concomitant disease(s) or any additional condition(s) which the investigator feels constitute(s) criteria for exclusion of a particular subject
* Major amputation required within 30 days
* Inclusion in any other clinical study that may affect the outcome of this study
* Uncorrected stenosis(es) of greater than 50% in the common and/or external iliac artery and/or common femoral artery of the index leg.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-06; Primary Completion 2016-06 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Murphy, MD, Principal Investigator — Indiana University School of Medicine
Locations (25):
- United States (25):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of California-Davis Medical Center, Sacramento, California
  - University of Miami, Miami, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - UMass Memorial Health Care, Worcester, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - Nebraska-Western Iowa VA Healthcare System, Omaha, Nebraska
  - Holy Name Medical Center, Teaneck, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - Weill Cornell Medical College / New York-Presbyterian Hospital, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Remington-Davis, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - University of Virginia Hospital, Charlottesville, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murphy MP, Lawson JH, Rapp BM, Dalsing MC, Klein J, Wilson MG, Hutchins GD, March KL. Autologous bone marrow mononuclear cell therapy is safe and promotes amputation-free survival in patients with critical limb ischemia. J Vasc Surg. 2011 Jun;53(6):1565-74.e1. doi: 10.1016/j.jvs.2011.01.074. Epub 2011 Apr 22. PMID 21514773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the study occurred between June 2010 and June 2015. Until February 2014, participants completing the initial 52-week follow-up period could choose to have their second limb randomized if the participant and limb continued to meet all study inclusion and exclusion criteria. Three (3) limbs were enrolled during this time, resulting in a total of 155 limbs in 152 participants that were included in the final intent-to treat analysis for the primary endpoint.
Pre-assignment Details: Participants that provided informed consent, completed all screening assessments, and met all inclusion and exclusion criteria for the study went on to be randomized and undergo the study procedure.
Units Other Than Participants: Limbs
Period: Overall Study
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
Started | 117; 119 Limbs | 36; 36 Limbs (One participant is counted in both treatment groups due to one leg being randomized to each group.)
Completed | 65; 67 Limbs | 19; 19 Limbs (Incl. 11 participants that received crossover treatment after completing 52 week primary follow up.)
Not Completed | 52; 52 Limbs | 17; 17 Limbs
Not completed — Met study endpoint (major amputation, death) | 36 | 16
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 6 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Received 2nd treatment via compassionate use | 1 | 0
Not completed — Early study termination by sponsor. | 2 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Limbs
Groups:
- Total: Total of all reporting groups
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham) | Total
Number analyzed (Participants) | 117 | 36 | 153
Number analyzed (Limbs) | 119 | 36 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age for all limbs. If a participant had multiple limbs evaluated, his/her age would be included multiple times in the analysis.
  years | 64.7 (11.9) | 66.7 (12.2) | 65.0 (11.9)
Sex: Female, Male [Count of Units; unit: Limbs]
  Female | 48 | 16 | 64
  Male | 71 | 20 | 91
Race/Ethnicity, Customized [Count of Units; unit: Limbs] — Count of race/ethnicity for all limbs. If a participant had multiple limbs evaluated, his/her race/ethnicity would be included multiple times in the analysis.
  Limbs
    African-American | 24 | 4 | 28
    White (non-Hispanic) | 91 | 27 | 118
    White (Hispanic) | 3 | 4 | 7
    Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 117 | 36 | 153
Rutherford Score [Count of Units; unit: Limbs] — The Rutherford score is a classification of severity for peripheral artery disease which ranges from 0 (asymptomatic) to 6 (major tissue loss extending above the transmetatarsal level, functional foot no longer salvageable). The study enrolled participants with Rutherford scores of 4 (ischemic rest pain) and 5 (minor tissue loss, nonhealing ulcer, and/or focal dry gangrene).
  Limbs
    Rutherford Score = 4 | 65 | 19 | 84
    Rutherford Score = 5 | 54 | 17 | 71
Diabetic Status [Count of Units; unit: Limbs] — Describes diabetic status of all limbs. If a participant had multiple limbs evaluated, his/her diabetic status would be included multiple times in the analysis.
  Limbs
    Diabetes = Yes | 49 | 14 | 63
    Diabetes = No | 70 | 22 | 92

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Major Amputation or Death
Description: Occurrence of major amputation (above the ankle joint) or death.
Time Frame: 52 weeks
Population: All limbs that were randomized to a treatment group were included in the analysis for the primary endpoint.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
Number analyzed (Participants) | 117 | 36
Number analyzed (Limbs) | 119 | 36
Limbs | 24 | 11
Statistical Analysis 1: Comparison: Concentrated Bone Marrow Aspirate (cBMA) vs Placebo Control (Sham); Test type: Superiority; p = 0.224, Proportional Hazards Regression; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.31 to 1.31]

2. Secondary Outcome: Visual Analog Scale (VAS) - Pain
Description: Pain reported at the 52-week follow-up visit as assessed on the visual analog scale (VAS). Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The distance from the beginning of the line is measured and reported in centimeters (cm), with 0 representing no pain and 10 representing the worst possible pain.
Time Frame: 52 weeks
Population: All limbs that were randomized to a treatment group, did not meet a primary endpoint or otherwise exit from the study, and that had an assessment available at 52 weeks were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Limbs
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
Number analyzed (Participants) | 117 | 36
Number analyzed (Limbs) | 119 | 36
score on a scale
  Baseline | 6.462 (7.789) | 5.836 (2.680)
  52 Weeks: number analyzed (Participants) | 94 | 24
  52 Weeks: number analyzed (Limbs) | 96 | 24
  52 Weeks | 3.651 (2.964) | 3.346 (3.019)
Statistical Analysis 1: Comparison: Concentrated Bone Marrow Aspirate (cBMA) vs Placebo Control (Sham); Test type: Superiority; p = 0.671, Repeated measures model — Treatment-by-week p-value is reported; The statistical analysis model includes treatment group, week, treatment-by-week, and baseline pain measurement

3. Secondary Outcome: Six-Minute Walk Test
Description: Measurement (in meters) of the total distance a participant is able to walk in 6 minutes. Since ability to walk is related to the condition of the affected limb, this measure is tied to limb pain and function. If a participant had multiple limbs included in the study, each limb was evaluated separately. Only one limb could be included in the study at a time.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters
Units Other Than Participants: Limbs
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
Number analyzed (Participants) | 117 | 36
Number analyzed (Limbs) | 119 | 36
meters
  Baseline: number analyzed (Participants) | 113 | 35
  Baseline: number analyzed (Limbs) | 115 | 35
  Baseline | 158.508 (115.157) | 173.114 (130.397)
  52 Weeks: number analyzed (Participants) | 82 | 23
  52 Weeks: number analyzed (Limbs) | 84 | 23
  52 Weeks | 223.545 (170.015) | 218.352 (148.226)
Statistical Analysis 1: Comparison: Concentrated Bone Marrow Aspirate (cBMA) vs Placebo Control (Sham); Test type: Superiority; p = 0.714, Repeated measures model — Treatment-by-week p-value is reported; The statistical analysis model includes treatment group, week, treatment-by-week, and baseline pain measurement

4. Other Pre Specified Outcome: Occurrence of Major Amputation or Death
Description: Occurrence of major amputation (above the ankle joint) or death for all participants through final follow-up.
Time Frame: 5 years
Population: All randomized participants were included in the analysis. Some participants did not re-consent for follow-up after 52 weeks and as such their long-term status is unknown. For the purposes of this analysis, they are counted with those who completed follow-up. Control participants that received crossover therapy with cBMA after 52 weeks are counted with the control group.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
Number analyzed (Participants) | 117 | 36
Number analyzed (Limbs) | 119 | 36
Limbs | 36 | 16

5. Post Hoc Outcome: Occurrence of Major Amputation or Death, Excluding Rutherford 5 Diabetic Subjects
Description: Occurrence of major amputation (above the ankle joint) or death, excluding the subgroup of subjects with Rutherford Category 5 critical limb ischemia and diabetes.
  The Rutherford score is a classification of severity for peripheral artery disease which ranges from 0 (asymptomatic) to 6 (major tissue loss extending above the transmetatarsal level, functional foot no longer salvageable). The study enrolled participants with Rutherford scores of 4 (ischemic rest pain) and 5 (minor tissue loss, nonhealing ulcer, and/or focal dry gangrene).
Time Frame: 52 weeks
Population: All limbs for subjects from the following subgroups that were randomized to a treatment group were included in this post-hoc analysis: Rutherford Category 4 and diabetic, Rutherford Category 4 and non-diabetic, Rutherford Category 5 and non-diabetic.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
Number analyzed (Participants) | 92 | 30
Number analyzed (Limbs) | 94 | 30
Limbs | 13 | 10
Statistical Analysis 1: Comparison: Concentrated Bone Marrow Aspirate (cBMA) vs Placebo Control (Sham); Test type: Superiority; p = 0.018, Proportional Hazards Regression; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.16 to 0.85]

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the start of study treatment up to the 52-week follow-up visit were recorded. Between 52 weeks and 5 years, only major adverse limb events, including those resulting in major amputation, and death were recorded. Serious adverse events are reported through 52 weeks. All-cause mortality is reported through 5 years. Not all participants re-consented to additional follow-up after week 52, so mortality information was only available for those that re-consented.
Description: Participants were asked to report adverse events during all follow-up visits, and site staff were to review medical records available between visits to determine if additional events had occurred that were not reported by participants. Although some events were not limb-related, they were recorded and counted for each enrolled limb. If a participant had multiple limbs included in the study, events for each limb were evaluated separately. Only one limb was included in the study at a time.
Arm/Group | Concentrated Bone Marrow Aspirate (cBMA) | Placebo Control (Sham)
All-Cause Mortality (participants affected / at risk) | 11/119 | 7/36
Serious Adverse Events (participants affected / at risk) | 66/119 | 24/36
Other Adverse Events (participants affected / at risk) | 117/119 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concentrated Bone Marrow Aspirate (cBMA) (N=119) | Placebo Control (Sham) (N=36)
Major Amputation - Index Leg (Surgical and medical procedures) | 19 | 8
Pain - Index Leg (Musculoskeletal and connective tissue disorders) | 7 | 6
Cellulitis - Index Leg (Infections and infestations) | 7 | 3
Death (General disorders) | 5 | 3
Ischemia - Index Leg (Vascular disorders) | 4 | 3
Toe Amputation - Index Leg (Surgical and medical procedures) | 5 | 2
Gangrene - Index Leg (Skin and subcutaneous tissue disorders) | 7 | 0
Pneumonia (Infections and infestations) | 6 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acute Congestive Heart Failure (Cardiac disorders) | 3 | 2
Wound - Index Leg (Skin and subcutaneous tissue disorders) | 5 | 1
Infection - Index Leg (Infections and infestations) | 4 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2
Bypass Graft - Index Leg (Surgical and medical procedures) | 1 | 2
Chest Pain (Cardiac disorders) | 3 | 3
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 | 2
Low Red Blood Cell-Related Level (Blood and lymphatic system disorders) | 2 | 1
Stroke (Vascular disorders) | 2 | 1
Osteomyelitis - Index Leg (Infections and infestations) | 4 | 0
Ulceration - Index Leg (Skin and subcutaneous tissue disorders) | 0 | 2
Sepsis (Infections and infestations) | 1 | 1
Wound - Contralateral Leg (Skin and subcutaneous tissue disorders) | 1 | 1
Ischemic Bowel (Gastrointestinal disorders) | 2 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (General disorders) | 2 | 0
Amputation of Foot - Contralateral Foot (Surgical and medical procedures) | 0 | 1
Amputation of Toe - Contralateral Leg (Surgical and medical procedures) | 0 | 1
Anaphylaxis Related to Antibiotic (Immune system disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hemorrhagic Anemia (Blood and lymphatic system disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Major Amputation - Contralateral Leg (Surgical and medical procedures) | 0 | 1
Non-ST-Elevation Myocardial Infarction (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
General Weakness (General disorders) | 0 | 1
Weakness - Hand (Metabolism and nutrition disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Abdominal Sepsis/Shock (Infections and infestations) | 1 | 0
Abscess - Buttock (Skin and subcutaneous tissue disorders) | 1 | 0
Angioplasty - Contralateral Leg (Surgical and medical procedures) | 1 | 0
Angioplasty - Index Leg (Surgical and medical procedures) | 1 | 0
Asystole Episode (Cardiac disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Decompensation (Cardiac disorders) | 1 | 0
Cardiac Ischemia (Vascular disorders) | 1 | 0
Carotid Blockage (Vascular disorders) | 1 | 0
Cellulitis - Arm (Infections and infestations) | 1 | 0
Cellulitis - Bilateral Legs (Infections and infestations) | 1 | 0
Cellulitis - Contralateral Leg (Infections and infestations) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Deep Vein Thrombosis - Index Leg (Vascular disorders) | 1 | 0
Deconditioning (Vascular disorders) | 1 | 0
Degenerative Disc - Cervical Spine (Musculoskeletal and connective tissue disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Elective Surgery (Surgical and medical procedures) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibroids (Reproductive system and breast disorders) | 1 | 0
Fracture - Contralateral Leg (Injury, poisoning and procedural complications) | 1 | 0
Hematoma (General disorders) | 1 | 0
Hyperglycemia (Investigations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Ileocolic Anastomotic Leak (Gastrointestinal disorders) | 1 | 0
Infected Abdominal Mesh (Infections and infestations) | 1 | 0
Infection - Contralateral Leg (Infections and infestations) | 1 | 0
Intra-Abdominal Abscess (Infections and infestations) | 1 | 0
Knee Revision - Index Leg (Surgical and medical procedures) | 1 | 0
Large Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Menstruation (Reproductive system and breast disorders) | 1 | 0
Metabolic Acidosis (Investigations) | 1 | 0
Near Syncope (Vascular disorders) | 1 | 0
Non-Healing of Toe Amputation Site (General disorders) | 1 | 0
Osteomyelitis - Contralateral Leg (Infections and infestations) | 1 | 0
Oversedation (Nervous system disorders) | 1 | 0
Pain - Contralateral Leg (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral Artery Disease (Vascular disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Prolonged Hospitalization (General disorders) | 1 | 0
Superior Mesenteric Artery Thrombus (Vascular disorders) | 1 | 0
Shortness of Breath (Cardiac disorders) | 1 | 0
Stenosis of Bypass Graft - Index Leg (Vascular disorders) | 1 | 0
Subarachnoid Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
Ulceration - Contralateral Leg (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Venous Thromboembolism - Contralateral Leg (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concentrated Bone Marrow Aspirate (cBMA) (N=119) | Placebo Control (Sham) (N=36)
Low Red Blood Cell-Related Level (Blood and lymphatic system disorders) | 87 | 13
Pain - Index Leg (Musculoskeletal and connective tissue disorders) | 62 | 22
Pain - Bilateral Iliac Crests (General disorders) | 30 | 4 — Pain from bone marrow aspiration procedure.
Ulceration - Index Leg (Skin and subcutaneous tissue disorders) | 17 | 8
Low White Blood Cell-Related Level (Blood and lymphatic system disorders) | 17 | 5
Cellulitis - Index Leg (Infections and infestations) | 14 | 4
Erythema - Index Leg (Skin and subcutaneous tissue disorders) | 9 | 5
Edema - Index Leg (Metabolism and nutrition disorders) | 12 | 2
High White Blood Cell-Related Level (Blood and lymphatic system disorders) | 11 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 8 | 4
Pain - Back (Musculoskeletal and connective tissue disorders) | 10 | 2
Wound - Index Leg (Skin and subcutaneous tissue disorders) | 15 | 7
Pneumonia (Infections and infestations) | 7 | 3
Gangrene - Index Leg (Skin and subcutaneous tissue disorders) | 9 | 1 — Dry gangrene
Infection - Index Leg (Infections and infestations) | 10 | 0
Respiratory Infection (Infections and infestations) | 4 | 3
High Red Blood Cell-Related Level (Blood and lymphatic system disorders) | 5 | 2
Urinary Tract Infection (Infections and infestations) | 5 | 2
Urinary Retention (Renal and urinary disorders) | 6 | 1
Fever (General disorders) | 2 | 4
Acute Congestive Heart Failure (Cardiac disorders) | 4 | 2
Acute Kidney Injury (Renal and urinary disorders) | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 0
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 2
Bypass Graft - Index Leg (Surgical and medical procedures) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Fissure - Index Leg (Skin and subcutaneous tissue disorders) | 1 | 2
Numbness - Index Leg (Nervous system disorders) | 1 | 2
Pain - Hip (Musculoskeletal and connective tissue disorders) | 1 | 2
Pruritis - Index Leg (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No